CLINICAL TRIAL: NCT05465135
Title: The Evaluation of the Effect of Dihydroartemisinin in Patients With Polycystic Ovary Syndrome
Brief Title: The Effect of Dihydroartemisinin in PCOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Xiaoying Li, Director, Shanghai Zhongshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2020-115R
Record Dates: First submitted 2022-07-10; First posted 2022-07-19 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — artenimol

STUDY DESIGN:
Intervention Model Description: 20 participants with PCOS receive dihydroartemisinin for 3 months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dihydroartemisinin Group (Experimental): The subjects take Dihydroartemisinin, 40mg tid for 12 weeks
  Interventions: Drug: Dihydroartemisinin

INTERVENTIONS:
Drug: Dihydroartemisinin — Dihydroartemisinin 40mg three times a day for 12 consecutive weeks.

SUMMARY:
Artemisinin has been widely used as a first-line antimalarial drug in routine clinical practice. In recent years, it has been reported that Artemisinin also has some significant anti-inflammatory, anti-tumor and immune-modulating effects. The investigators' previous studies discovered that Artemisinin dramatically reduced serum androgen levels and improved poly-cystic ovary syndrome(PCOS) in animals. Preliminary study by the investigators found that artemisinin derivatives are capable of reducing both androgen levels and improving insulin resistance, two clinical characteristics of PCOS. Thus artemisinin derivatives has the potential effect to alleviate PCOS symptoms. The current study aims to investigate the effect of artemisinin on improving PCOS and serum androgen levels in PCOS subjects.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is a common reproductive endocrine metabolic disorder caused by a combination of genetic and environmental factors. The pathogenesis of PCOS remains unclear. Artemisinin has been widely used as a first-line antimalarial drug in routine clinical practice. In recent years, it has been reported that Artemisinin has significant anti-inflammatory, anti-tumor and immune-modulating effects. The investigator's previous studies found that artemisinin and its derivatives could significantly promote uncoupling protein 1 (UCP1) transcription and the conversion of white fat to brown fat. Artemisinin derivatives upregulated the levels of genes critical for brown fat differentiation and function, accompanied by enhanced mitochondrial biosynthesis, demonstrating their potential to promote white fat browning and improve metabolism in rodent models. The investigators also observed that androgen levels in drug-induced PCOS rats were reduced, when treated with artemether analogs for prophylactic and therapeutic purposes, respectively. It is believed that the two core mechanisms in the pathogenesis of PCOS are excessive androgen synthesis and insulin resistance. Preliminary study by the investigators found that artemisinin derivatives are capable of reducing both serum androgen levels and improving insulin resistance, two clinical characteristics of PCOS. Thus artemisinin derivatives has the potential effect to alleviate PCOS symptoms and control or even reverse the disease progression. The current study aims to investigate the effect of artemisinin on improving PCOS and serum androgen levels in PCOS subjects.

ELIGIBILITY:
Inclusion Criteria:

* BMI 23-30kg/M2
* No plan for pregnancy in the coming 6 months
* Newly diagnosed PCOS, or PCOS without any medication for the past three months.
* Patients should meet all the three following criteria:

  1. Oligomenorrhea or amenorrhea: Oligomenorrhea is defined as more than 35 days between menstrual periods and less than 8 menstrual bleedings in the past year; amenorrhea is defined as more than 90 days between two menstrual bleedings.
  2. Polycystic ovaries: ≥12 follicles in both ovaries (diameter<10mm), confirmed by ultrasound.
  3. Elevated androgen levels: testosterone>1.67 nmol/L.

Exclusion Criteria:

* Previously treated with steroids or other medications for PCOS in the past 3 months.
* Patients with other endocrine diseases that can cause secondary PCOS, including but not limited to: 21 hydroxylase deficiency, prolactinoma, hypothyroidism, Cushing's syndrome, etc.
* Pregnancy.
* Patients with other serious diseases affecting heart, liver, kidney, or other major organs.
* Patients with any type of cancer.

Ages: 16 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-04-23 (Actual)

PRIMARY OUTCOMES:
Recovery of regular menses by questionnaire | 12 weeks
  Periodical vaginal bleeding by questionnaire
Bilateral ovary volume | 12 weeks
  Length, width and height of bilateral ovaries measured by B type ultrasound
Number of immature follicles | 12 weeks
  Total number of follicles with diameters <10 mm measured by B type ultrasound
Serum testosterone levels | 12 weeks
  Measurement of serum total testosterone

SECONDARY OUTCOMES:
Serum anti-Mullerian hormone | 12 weeks
  Measurement of serum AMH
Sex hormone binding globulin (SHBG) | 12 weeks
  Measurement of serum SHBG
Serum dehydroepiandrosterone sulfate | 12 weeks after drug intervention
  Measurement of serum DHEA

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoying Li, MD, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No